CLINICAL TRIAL: NCT01099930
Title: Targeting Multiple Sclerosis as an Autoimmune Disease With Intensive Immunoablative Therapy and Immunological Reconstitution: A Potential Curative Therapy for Patients With a Predicted Poor Prognosis
Brief Title: Autologous Stem Cell Transplant for Multiple Sclerosis
Acronym: MS/BMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Multiple Sclerosis Scientific Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200037401H
Record Dates: First submitted 2010-03-01; First posted 2010-04-08 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
Keywords: immunoablation; stem cell transplantation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-randomized control group (Active Comparator): Patients meeting inclusion/exclusion criteria not consenting to treatment will be requested to consent to control group and followed while receiving standard of care.
  Interventions: Other: Standard Therapy
- Stem Cell Transplantation (Experimental): Patients will undergo stem cell transplantation for the treatment of Multiple Sclerosis
  Interventions: Other: immuno-ablation and autologous CD34 selected hematopoietic stem cell transplantation (HSCT),

INTERVENTIONS:
Other: immuno-ablation and autologous CD34 selected hematopoietic stem cell transplantation (HSCT), — Stem Cell Mobilization with Cyclophosphamide 4.5 gm/m2 and rhGCSF 10 ug/kg/d x 10 day.
  Stem Cell Collection with Cobe Spectra Stem Cell Purification with Miltenyi CliniMACS Stem Cell Transplant Conditioning with Busulphan 9.6 mg/kg iv, Cyclophosphamide 200 mg/kg iv, rabbit ATG 5 mg/kg iv followed by CD34 selected autologous hematopoietic stem cell transplant
  Arms: Stem Cell Transplantation
Other: Standard Therapy — Patient will receive standard therapy as decided upon by their treating neurologist.
  Arms: Non-randomized control group

SUMMARY:
Multiple sclerosis is an autoimmune disease. We are studying whether high dose chemotherapy and autologous stem cell transplant can replace the autoreactive immune system and if this reduces clinical inflammatory disease in the central nervous system (CNS). A second goal is to examine whether there is long-term stabilization or improvement in disability scores if the inflammatory disease is controlled.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* The diagnosis of active multiple sclerosis with relapses or progression and sustained accumulated impairment, made by a neurologist expert in the field
* Patient considered at high risk of progression
* EDSS Cerebellar Functional score greater than or equal to 3 OR EDSS Pyramidal Functional score greater than or equal to 3
* EDSS between greater than or equal to 3 and less than or equal to 6
* Evidence of current disease activity
* Evidence of progression or continued relapses or worsening MRI after at least one year of therapy with interferon-B1, glatiramer acetate, Mitoxantrone, or other conventional dose immunosuppressive drug therapy
* If a patient has previously received a cytotoxic agent (Mitoxantrone, Cyclophosphamide etc.) they must have normal bone marrow morphology and cytogenetics before being considered eligible for this study
* MRI brain scan that satisfies the MRI criteria of Paty or Fazekas for the diagnosis of multiple sclerosis
* No evidence of hepatic inflammation or fibrosis

Exclusion Criteria:

* Patients with primary progressive multiple sclerosis
* Patients with cardiac, renal, pulmonary, hepatic or other organ impairment that would limit their ability to receive dose intensive immunosuppressive therapy including high dose chemotherapy and ASCT
* Patient with any active or chronic infection
* Patients who are seropositive for HIV1, HIV2, Hepatitis B Surface Antigen, and Hepatitis C
* Patients with a previous history of a malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
* Patients whose life expectancy is severely limited by another co-morbid illness
* Patients with evidence of myelodysplasia or other non-autoimmune cytopenia
* Patients having received a cytotoxic agent within one month of enrolling in this study
* Pregnancy or risk of pregnancy. This includes patients that are unwilling to practice active contraception during the time of chemotherapy
* Patients with hypersensitivity to rabbit proteins
* Patients unable to give written informed consent in accordance with research ethics board guidelines
* Patients having previous exposure to natalizumab or alemtuzumab.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2001-08; Primary Completion 2012-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
3 year MS activity free survival | 3 year follow-up post transplant

SECONDARY OUTCOMES:
Transplant related morbidity | 3 year follow-up post transplant
Transplant related mortality | 3 years
Time to MS treatment failure | 3 years
rate of immune reconstitution following treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harold L Atkins, MD, Principal Investigator — Ottawa Hospital Research Institute; Mark S Freedman, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Atkins HL, Bowman M, Allan D, Anstee G, Arnold DL, Bar-Or A, Bence-Bruckler I, Birch P, Bredeson C, Chen J, Fergusson D, Halpenny M, Hamelin L, Huebsch L, Hutton B, Laneuville P, Lapierre Y, Lee H, Martin L, McDiarmid S, O'Connor P, Ramsay T, Sabloff M, Walker L, Freedman MS. Immunoablation and autologous haemopoietic stem-cell transplantation for aggressive multiple sclerosis: a multicentre single-group phase 2 trial. Lancet. 2016 Aug 6;388(10044):576-85. doi: 10.1016/S0140-6736(16)30169-6. Epub 2016 Jun 9. PMID 27291994
- [Derived] Bose G, Atkins HL, Bowman M, Freedman MS. Autologous hematopoietic stem cell transplantation improves fatigue in multiple sclerosis. Mult Scler. 2019 Nov;25(13):1764-1772. doi: 10.1177/1352458518802544. Epub 2018 Sep 25. PMID 30251913
- [Derived] Darlington PJ, Stopnicki B, Touil T, Doucet JS, Fawaz L, Roberts ME, Boivin MN, Arbour N, Freedman MS, Atkins HL, Bar-Or A. Natural Killer Cells Regulate Th17 Cells After Autologous Hematopoietic Stem Cell Transplantation for Relapsing Remitting Multiple Sclerosis. Front Immunol. 2018 May 7;9:834. doi: 10.3389/fimmu.2018.00834. eCollection 2018. PMID 29867923